CLINICAL TRIAL: NCT04486261
Title: High-intensity Strength Training in Patients With Idiopathic Inflammatory Myopathies: Changes in Quality of Life, Muscle Strength, Function and Myocellular Parameters
Brief Title: High-intensity Strength Training in Myositis
Acronym: HI-STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Southern Denmark (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Louise Pyndt Diederichsen, Consultant Rheumatologist, Associate professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCT16072020
Record Dates: First submitted 2020-07-17; First posted 2020-07-24 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Myositis; Dermatomyositis; Polymyositis; Immune-Mediated Necrotizing Myopathy
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity strength training (Experimental): 16 weeks of high-intensity strength training two times per week.
  Participants will receive the usual care in accordance to myositis (various DMARDs, different from patient to patient)
  Interventions:
  Other: high-intensity strength training Drug: Usual care
  Interventions: Other: High-intensity strength training
- Control (No Intervention): Participants receive the usual care in accordance to myositis (various DMARDs, different from patient to patient).
  Intervention:
  Drug: Usual care

INTERVENTIONS:
Other: High-intensity strength training — The high-intensity strength training protocol will consist of 2 training sessions per week. The first two weeks will be familiarisation training, where each exercise will be performed in three sets of 10 repetitions at an intensity of 15 repetitions maximum (RM). At week three each session will consist of 3 sets of each exercise corresponding to 10 RM, which will be kept for the remaining part of training intervention. The weights for each exercise will be adjusted throughout the intervention period, so the training load will correspond to 10 RM for each exercise in the entire intervention period.
  Other Names: High-intensity resistance training
  Arms: High-intensity strength training

SUMMARY:
This study evaluates the effects of a high-intensity strength training in patients with myositis with the primary outcome being quality of life (SF-36). The study is designed as a parallel group randomised controlled trial with an intervention group and a control group.

DETAILED DESCRIPTION:
Overall aim:

To investigate the effect of high-intensity strength training on quality of life, muscle strength, physical function, and disease activity in patients with myositis

Study design:

60 myositis patients will be included in a 16-week high-intensity strength training study. Patients will be randomly allocated into 2 groups (strength training and control) in a 1:1 ratio.

User involvement:

Myositis patients has been recruited to a patient advisory board. The advisory board's objective is to give patient-oriented project feedback, thus improving the overall research project.

Intervention:

Two training session per week for 16 weeks. Sessions consists of 3 sets of each exercise corresponding to 10 RM. Training progression will be accounted for and training loads will be evaluated weekly. The training protocol will be a full-body protocol, i.e. all major muscle groups will be engaged during each training session.

Outcomes:

The primary outcome is the Physical Component Summary Measure from the quality of life questionnaire (SF-36). Secondary outcomes include strength measures, functional tests, disease activity measures, questionnaires (e.g. International physical activity questionnaire), DEXA whole body scans, blood samples and muscle biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the criteria for myositis by EULAR/ACR (Bottai et al., 2017; Lundberg et al., 2017)
* ≤ 5 mg/day Prednisolone
* Stable dosage of immunosuppressive treatment for at least 1 months prior to inclusion in the study
* Myositis diagnosis at least 6 months prior to inclusion in the study

Exclusion Criteria:

* Patients with sporadic inclusion body myositis and overlap myositis (myositis combined with another autoimmune rheumatic diseases, except Sjögren's Syndrome)
* Co-morbidity preventing resistance training (severe heart/lung-disease, uncontrolled hypertension (systolic > 160mmHg, diastolic > 100mmHg), severe knee/hip arthritis)
* Alcohol- and/or drug abuse. Defined by the guidelines issued by The Danish Health Authority

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Quality of life (health survey (SF-36) subscale: Physical Component Summary) | 16 weeks
  Quality of life will be evaluated with the short form (36) health survey (SF-36) subscale: Physical Component Summary. The scale ranges from 0 to 100 where 100 is the highest score.

SECONDARY OUTCOMES:
Leg power | 16 weeks
  Power rig
Handgrip strength | 16 weeks
  Measured by a handheld dynamometer
Functional Index 3 | 16 weeks
  A test of muscle strength in a series of muscles, carried out by the physician or physiotherapist
30 seconds chair rise | 16 weeks
  Participants are instructed to stand up and sit down on a chair as many times as possible in 30 sec.
Timed up-and-go | 16 weeks
  Participants are instructed to rise from a chair walk 3 m forward, pass a marking and return to the chair and sit down as fast as possible
2-minute walk test | 16 weeks
  A 2-min maximal walk test where the participant is encouraged to cover the greatest distance possible.
Balance | 16 weeks
  Short physical performance battery - balance part
Whole-body, appendicular and lower-limb lean mass | 16 weeks
  Measured by Dual-energy X-ray absorptiometry
Fat-free mass, body fat and total mass | 16 weeks
  Measured by bioimpedance
Physician Global Activity | 16 weeks
  Physician's overall assessment on a single 0-10 cm scale, where the higher score indicates higher disease activity
Patient Global Activity | 16 weeks
  Patient's overall assessment on a single 0-10 cm scale, where the higher score indicates higher disease activity.
Extra-muscular Disease Activity | 16 weeks
  An assessment tool used by the physician to evaluate disease activity in various organ systems via a scoring system and a 0-10 cm scale, where the higher score indicates higher disease activity.
Manual muscle test 8 | 16 weeks
  A test of muscle strength in a series of muscles, carried out by the physician
Health Assessment Questionnaire (HAQ) | 16 weeks
  HAQ is a questionnaire to evaluate patient reported disability. It has 8 categories with a range of questions. Each question is scored from 0 to 3 where 0 is no disability and 3 is unable to do.
Physician Global assessment of disease damage | 16 weeks
  Physician's overall assessment on a single 0-10 cm scale, where the higher score indicates higher disease damage.
Patient Global assessment of disease damage | 16 weeks
  Patient's overall assessment on a single 0-10 cm scale, where the higher score indicates higher disease damage.
Medical history | 16 weeks
  Questionnaire:
  Basic cardiovascular questionnaire concerning medical conditions, current medication, heart symptoms and smoking habits
Self-perceived physical activity levels | 16 weeks
  International Physical Activity Questionnaire - long
Quality of life (health survey (SF-36) subscale: Mental component summary) | 16 weeks
  Quality of life will be evaluated with the short form (36) health survey (SF-36) subscale: Mental Component Summary. The scale ranges from 0 to 100 where 100 is the highest score.
Body mass index (BMI) | 16 weeks
  Weight will be measured by scale (kg). Height will be measured by measuring (m). BMI will be derived from weight and height (kg/m^2)
Systolic and diastolic blood pressure | 16 weeks
  Measured by blood pressure monitor
Blood samples (analysis of markers of af disease activity) | 16 weeks
  Plasma analysis: lipid profile, HbA1c, troponins, NT-proBNP, creatine kinase
Electrocardiography (ECG) | 16 weeks
  Standard 12-lead ECG at 25 mm/s is recorded and analyzed according to standard published criteria (48-50). According to the Minnesota coding the PQ-interval is measured and presence of 1st, 2nd (including Mobitz type 1 and 2), and 3rd degree of AV block are noted. Additional measures will include: P-wave duration (≥ 2.5 mm in any of leads II, III, aVF), QRS duration (≥ 120 ms in any of leads I, II, III, aVL, aVF), QTc duration (> 450 ms), atrial fibrillation and flutter.

OTHER OUTCOMES:
Muscle biopsies | 16 weeks
  Muscle biopsies will be taken on a selected number of subjects from either the vastus lateralis or the tibialis anterior muscle, for the use in future analysis of i.e. muscle fibre size and distribution, myogenic stem cell activity, capillary density, muscle inflammation ect.
Physical activity level | 16 weeks
  Will be measured by activity tracker (watch)

CONTACTS AND LOCATIONS:
Overall Officials: Louise Pyndt Diederichsen, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to GDPR-regulations IPD will not be available.

REFERENCES:
- [Background] Bottai M, Tjarnlund A, Santoni G, Werth VP, Pilkington C, de Visser M, Alfredsson L, Amato AA, Barohn RJ, Liang MH, Singh JA, Aggarwal R, Arnardottir S, Chinoy H, Cooper RG, Danko K, Dimachkie MM, Feldman BM, Garcia-De La Torre I, Gordon P, Hayashi T, Katz JD, Kohsaka H, Lachenbruch PA, Lang BA, Li Y, Oddis CV, Olesinka M, Reed AM, Rutkowska-Sak L, Sanner H, Selva-O'Callaghan A, Wook Song Y, Vencovsky J, Ytterberg SR, Miller FW, Rider LG, Lundberg IE; International Myositis Classification Criteria Project consortium, the Euromyositis register and the Juvenile Dermatomyositis Cohort Biomarker Study and Repository (JDRG) (UK and Ireland). EULAR/ACR classification criteria for adult and juvenile idiopathic inflammatory myopathies and their major subgroups: a methodology report. RMD Open. 2017 Nov 14;3(2):e000507. doi: 10.1136/rmdopen-2017-000507. eCollection 2017. PMID 29177080
- [Background] Lundberg IE, Tjarnlund A, Bottai M, Werth VP, Pilkington C, de Visser M, Alfredsson L, Amato AA, Barohn RJ, Liang MH, Singh JA, Aggarwal R, Arnardottir S, Chinoy H, Cooper RG, Danko K, Dimachkie MM, Feldman BM, Garcia-De La Torre I, Gordon P, Hayashi T, Katz JD, Kohsaka H, Lachenbruch PA, Lang BA, Li Y, Oddis CV, Olesinska M, Reed AM, Rutkowska-Sak L, Sanner H, Selva-O'Callaghan A, Song YW, Vencovsky J, Ytterberg SR, Miller FW, Rider LG; International Myositis Classification Criteria Project Consortium, the Euromyositis Register, and the Juvenile Dermatomyositis Cohort Biomarker Study and Repository (UK and Ireland). 2017 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Adult and Juvenile Idiopathic Inflammatory Myopathies and Their Major Subgroups. Arthritis Rheumatol. 2017 Dec;69(12):2271-2282. doi: 10.1002/art.40320. Epub 2017 Oct 27. PMID 29106061
- [Derived] Jensen KY, Aagaard P, Suetta C, Nielsen JL, Bech RD, Schroder HD, Christensen J, Simonsen C, Diederichsen LP. High-intensity resistance training in patients with myositis - 1-year follow-up on a randomised controlled trial. Rheumatol Int. 2025 Apr 16;45(5):104. doi: 10.1007/s00296-025-05858-8. PMID 40237840
- [Derived] Jensen KY, Aagaard P, Suetta C, Nielsen JL, Bech RD, Schroder HD, Christensen J, Simonsen C, Diederichsen LP. High-intensity resistance training improves quality of life, muscle endurance and strength in patients with myositis: a randomised controlled trial. Rheumatol Int. 2024 Oct;44(10):1909-1921. doi: 10.1007/s00296-024-05698-y. Epub 2024 Aug 27. PMID 39192022
- [Derived] Jensen KY, Aagaard P, Schroder HD, Suetta C, Nielsen JL, Boyle E, Diederichsen LP. High-intensity strength training in patients with idiopathic inflammatory myopathies: a randomised controlled trial protocol. BMJ Open. 2021 Jun 25;11(6):e043793. doi: 10.1136/bmjopen-2020-043793. PMID 34172544